CLINICAL TRIAL: NCT00461786
Title: A Phase II Evaluation of Pemetrexed (Alimta, LY231514l, IND # 40061) in the Treatment of Recurrent or Persistent Platinum Resistant Ovarian or Primary Peritoneal Carcinoma
Brief Title: A Study of Single Agent Pemetrexed Disodium in Treating Patients With Recurrent or Persistent Ovarian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8364; H3E-US-JMGP
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2009-08-24 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Ovarian Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed (Experimental)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 900 mg/m2, intravenous (IV), every 21 days, until disease progression
  Other Names: LY231514; Alimta

SUMMARY:
The primary purpose of this trial is to estimate the drug effect on tumors in patients with ovarian or primary peritoneal cancers. Patients will receive Pemetrexed every 21 days until disease progression or unacceptable toxicity. This medication will be given over 10 minutes and may be administered intravenously (IV), through a vein in your arm. Vitamin supplementation is a required part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or persistent disease ovarian epithelial or primary peritoneal cancer
* Measurable disease
* Must have received 1 prior platinum-based (carboplatin, cisplatin, or another organoplatinum compound) chemotherapy regimen for primary disease. Patients who had not received prior paclitaxel may have received a second regimen that included paclitaxel
* Treatment-free interval < 6 months after prior platinum-based therapy OR progressed during platinum-based therapy
* Not eligible for a higher priority Gynecologic Oncology Group (GOG) protocol (i.e., any active phase III GOG protocol for the same patient population)

Exclusion Criteria:

* Patients who have had prior therapy with pemetrexed
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients who have received radiation to more than 25% of marrow

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed: Pemetrexed 900 mg/m2, intravenous (IV), every 21 days, until disease progression
Period: Overall Study
Arm/Group | Pemetrexed
Started | 51
Completed | 48 (Completed means the patient was evaluable for response.)
Not Completed | 3
Not completed — Entry Criteria Not Met | 2
Not completed — Inevaluable (Never Treated) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 48
Age, Customized [Number; unit: participants]
  <40 years | 1
  40-49 years | 6
  50-59 years | 14
  60-69 years | 14
  70-79 years | 11
  >79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 48
Cell Type [Number; unit: participants]
  Serous | 34
  Clear Cell | 5
  Mixed Epithelial | 6
  Endometrioid | 1
  Adenocarcinoma, Unspecified | 1
  Undifferentiated Carcinoma | 1
Gynecologic Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully active | 30
    1 - Ambulatory, Restricted Strenuous Activity | 15
    2 - Ambulatory, No Work Activities | 3
Prior Chemotherapy [Number; unit: participants]
  Yes | 48
  No | 0
Prior Radiotherapy [Number; unit: participants]
  Yes | 1
  No | 47
Race/Ethnicity [Number; unit: participants]
  White | 47
  Black | 1
Tumor Grade [Number; unit: participants] — Tumor grade is a system used to classify tumors based on certain characteristics of their cells. The grade is directly related to prognosis. The more they look like normal cells, the better the prognosis. Grades range from 1 (well-differentiated) to 4 (undifferentiated). The higher the grade, the worse the prognosis.
  participants
    1 - Well-Differentiated | 1
    2 - Moderately Differentiated | 15
    3 - Poorly Differentiated | 31
    Unspecified | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment. Complete response (CR) = disappearance of all target lesions; Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions; Stable disease (SD) = small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (up to 44 months)
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 48
participants
  Complete Response | 1
  Partial Response | 9
  Stable Disease | 17
  Progressive Disease | 18
  Inevaluable | 3
Statistical Analysis 1: Comparison: Pemetrexed; Overall Response Rate is the total percentage of participants with either a complete response or a partial response (CR+PR)/48 X 100; Test type: Superiority or Other; Overall Response Rate = 21, 95% CI [10.5 to 35.0]

2. Secondary Outcome: Number of Participants With Adverse Events by Grade
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) for defining and grading specific adverse events. A grading (severity) scale is provided for each adverse event term. Grades range from 0 (none) to 5 (death). The worst grade event per cycle is reported.
Time Frame: every 21-day cycle up to 5 year follow-up
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 48
participants
  Leukopenia - Grade 1 | 11
  Leukopenia - Grade 2 | 13
  Leukopenia - Grade 3 | 11
  Leukopenia - Grade 4 | 1
  Thrombocytopenia - Grade 1 | 15
  Thrombocytopenia - Grade 2 | 5
  Thrombocytopenia - Grade 3 | 2
  Thrombocytopenia - Grade 4 | 4
  Neutropenia - Grade 1 | 9
  Neutropenia - Grade 2 | 6
  Neutropenia - Grade 3 | 11
  Neutropenia - Grade 4 | 9
  Anemia - Grade 1 | 14
  Anemia - Grade 2 | 17
  Anemia - Grade 3 | 7
  Anemia - Grade 4 | 0
  Transfusion - Grade 1 | 0
  Transfusion - Grade 2 | 1
  Transfusion - Grade 3 | 0
  Transfusion - Grade 4 | 0
  Coagulation - Grade 1 | 0
  Coagulation - Grade 2 | 1
  Coagulation - Grade 3 | 0
  Coagulation - Grade 4 | 0
  Gastrointestinal - Grade 1 | 14
  Gastrointestinal - Grade 2 | 14
  Gastrointestinal - Grade 3 | 4
  Gastrointestinal - Grade 4 | 0
  Nausea/vomiting - Grade 1 | 15
  Nausea/vomiting - Grade 2 | 7
  Nausea/vomiting - Grade 3 | 4
  Nausea/vomiting - Grade 4 | 0
  Genitourinary - Grade 1 | 4
  Genitourinary - Grade 2 | 0
  Genitourinary - Grade 3 | 2
  Genitourinary - Grade 4 | 0
  Hepatic - Grade 1 | 2
  Hepatic - Grade 2 | 2
  Hepatic - Grade 3 | 1
  Hepatic - Grade 4 | 0
  Alopecia - Grade 1 | 7
  Alopecia - Grade 2 | 5
  Dermatologic - Grade 1 | 10
  Dermatologic - Grade 2 | 10
  Dermatologic - Grade 3 | 3
  Dermatologic - Grade 4 | 0
  Neurologic - Grade 1 | 12
  Neurologic - Grade 2 | 1
  Neurologic - Grade 3 | 4
  Neurologic - Grade 4 | 1
  SGOT - Grade 1 | 9
  SGOT - Grade 2 | 4
  SGOT - Grade 3 | 0
  SGOT - Grade 4 | 0
  Alkaline phosphatase - Grade 1 | 3
  Alkaline phosphatase - Grade 2 | 3
  Alkaline phosphatase - Grade 3 | 0
  Alkaline phosphatase - Grade 4 | 0
  Ocular - Grade 1 | 2
  Ocular - Grade 2 | 3
  Ocular - Grade 3 | 1
  Ocular - Grade 4 | 0
  Hemorrhage - Grade 1 | 2
  Hemorrhage - Grade 2 | 0
  Hemorrhage - Grade 3 | 1
  Hemorrhage - Grade 4 | 0
  Pulmonary - Grade 1 | 4
  Pulmonary - Grade 2 | 1
  Pulmonary - Grade 3 | 0
  Pulmonary - Grade 4 | 0
  Lymphopenia - Grade 1 | 1
  Lymphopenia - Grade 2 | 0
  Lymphopenia - Grade 3 | 0
  Lymphopenia - Grade 4 | 0
  Constitutional - Grade 1 | 17
  Constitutional - Grade 2 | 14
  Constitutional - Grade 3 | 5
  Constitutional - Grade 4 | 2
  Metabolic - Grade 1 | 20
  Metabolic - Grade 2 | 9
  Metabolic - Grade 3 | 4
  Metabolic - Grade 4 | 0
  Cardiovascular - Grade 1 | 3
  Cardiovascular - Grade 2 | 0
  Cardiovascular - Grade 3 | 0
  Cardiovascular - Grade 4 | 0
  Pain - Grade 1 | 8
  Pain - Grade 2 | 6
  Pain - Grade 3 | 1
  Pain - Grade 4 | 1
  Infection - Grade 1 | 2
  Infection - Grade 2 | 5
  Infection - Grade 3 | 5
  Infection - Grade 4 | 0
  Auditory - Grade 1 | 0
  Auditory - Grade 2 | 2
  Auditory - Grade 3 | 1
  Auditory - Grade 4 | 0
  Lymphatics - Grade 1 | 4
  Lymphatics - Grade 2 | 1
  Lymphatics - Grade 3 | 0
  Lymphatics - Grade 4 | 1
  Endocrine - Grade 1 | 2
  Endocrine - Grade 2 | 0
  Endocrine - Grade 3 | 0
  Endocrine - Grade 4 | 0
  Allergy - Grade 1 | 0
  Allergy - Grade 2 | 1
  Allergy - Grade 3 | 0
  Allergy - Grade 4 | 0

3. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: time of initial response until documented tumor progression (up to 44 months)
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 48
months | 8.4 [2.8 to 30.4]

4. Secondary Outcome: Progression-Free Survival
Description: Defined as the time from date of first dose to the first observation of disease progression, or death due to any cause.
Time Frame: baseline until documented tumor progression (up to 44 months)
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 48
months | 3.0 [1.0 to 33.1]

5. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline until death from any cause up to 5-year follow-up
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 48
months | 11.4 [1.6 to 34.4]

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 12/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (4)
Asthenia (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatinine abnormal (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed (N=48)
Anemia (Blood and lymphatic system disorders) | 38
Leukopenia (Blood and lymphatic system disorders) | 36
Lymphatics (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 35
Thrombocytopenia (Blood and lymphatic system disorders) | 26
Cardiovascular (Cardiac disorders) | 3
Auditory (Ear and labyrinth disorders) | 3
Ocular (Eye disorders) | 6
Gastrointestinal (Gastrointestinal disorders) | 32
Nausea/vomiting (Gastrointestinal disorders) | 26
Constitutional (General disorders) | 38
Pain (General disorders) | 16
Hepatic (Hepatobiliary disorders) | 5
Infection (Infections and infestations) | 12
Alkaline phosphatase (Investigations) | 6
Serum glutamic oxaloacetic transaminase (Investigations) | 13
Metabolic (Metabolism and nutrition disorders) | 33
Neurologic (Nervous system disorders) | 18
Genitourinary (Renal and urinary disorders) | 6
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 12
Dermatologic (Skin and subcutaneous tissue disorders) | 23
Hemorrhage (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days